CLINICAL TRIAL: NCT05517915
Title: Effect of Interval Inspiratory Muscle Training on Autonomic Dysfunction and Blood Pressure in Hypertensive Adults: A Randomized Controlled Trial
Brief Title: Inspiratory Muscle Training, Autonomic Dysfunction and Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Masood Khan, Principal Investigator, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16/9/139/JMI/IEC/2017
Record Dates: First submitted 2022-08-24; First posted 2022-08-26 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Hypertension
Keywords: Interval Inspiratory Muscle Training; Hypertension; Autonomic Dysfunction; Blood Pressure
MeSH Terms: conditions — Hypertension; Primary Dysautonomias

STUDY DESIGN:
Intervention Model Description: Two group pretest-posttest parallel design.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor was kept blind to the allocation of participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IMT group (Experimental): IMT training with 70% threshold was given.
  Interventions: Other: Inspiratory muscle training.
- Sham group (Sham Comparator): unloaded IMT training was given.
  Interventions: Other: Sham inspiratory muscle training.

INTERVENTIONS:
Other: Inspiratory muscle training. — Interval inspiratory muscle training was performed using the inspiratory muscle trainer.
  Arms: IMT group
Other: Sham inspiratory muscle training. — Interval inspiratory muscle training was performed using the unloaded inspiratory muscle trainer.
  Arms: Sham group

SUMMARY:
This study finds the effectiveness of inspiratory muscle threshold loading training among adults with hypertension. A sample of hypertensive subjects was divided into two groups - inspiratory muscle training (IMT) - group (inspiratory muscle training was prescribed) and sham-group (no load was prescribed during IMT). Both groups had training sessions comprising seven cycles of two minutes bouts of breathing counter to an inspiratory load, each bout parted by one minute of unloaded recovery. Treatment session was performed for three times per week for a total of six weeks. Measurement of each of the variables (blood pressure, resting heart rate (RHR), heart rate variability (HRV)) was taken at baseline and after the six-week intervention.

DETAILED DESCRIPTION:
The present study aimed to examine the outcome of interval inspiratory muscle training at 70% load on blood pressure, resting heart rate and autonomic dysfunction in the hypertensive adults.

Participants were divided into two groups: IMT and sham. In IMT group, the threshold loading inspiratory muscle trainer from POWERbreathe was used with 70% IMT threshold. In Sham group, IMT was unloaded.

ELIGIBILITY:
Inclusion Criteria:

* stage 1 hypertension
* essential hypertension
* mild hypertension

Exclusion Criteria:

* Subjects participating in exercise training for more than the last six months
* severe musculoskeletal limitations
* severe neurological limitations
* cognitive impairments
* uncontrolled diabetes
* uncontrolled hypertension
* a history of myocardial infarction (MI)
* a history of stroke in the last six months
* unstable angina
* chronic heart failure
* pulmonary disease of any etiology

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2018-06-18 (Actual); Study Completion 2018-08-27 (Actual)

PRIMARY OUTCOMES:
Resting heart rate | 6 weeks
  Resting heart rate was measured at baseline and after completion of intervention.
Autonomic functions | 6 weeks
  Autonomic functions were assessed by measuring the heart rate variability parameters at baseline and after completion of intervention.
Blood pressure | 6 weeks
  Systolic and diastolic blood pressures were measured at baseline and after completion of intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Masood Khan, M.P.Th, Principal Investigator — King Saud University
Locations (1):
- King Saud University, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No